CLINICAL TRIAL: NCT03099434
Title: Expanding Live Donor Kidney Transplantation Through Advocacy Training and Social Media
Acronym: ENGAGE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Alabama at Birmingham (Other); Northwestern University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: IRB00125128; R01DK111966 (NIH)
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Kidney Failure; Kidney Diseases
Keywords: Live Donor Transplant, Social Media, Education, Advocacy, Live Donor
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to one of the 3 arms, where arm 1 is two interventions combined (LDC program + Facebook app), arm 2 is one intervention (Facebook app), and arm 3 is the control group (standard-of-care).
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Live Donor Champion + Facebook App (Active Comparator): The LDC program consists of 6 monthly sessions of approx. 1 hour each. Each LDC session is led by a transplant physician or clinical coordinator. LDC sessions incorporate formal didactics, active-participant learning, personal stories, moderated group discussions, role-playing, and other skill-building exercises. LDC sessions are as follows: 1) education about ESRD, KT, and LDKT 2) communication skills building 3) Exploring social networks 4) sharing successful donor and recipient stories 5) encouraging candidate self-efficacy. At session 3, the the Facebook app will be incorporated and given to candidates. The Facebook app provides step-by-step instructions for creating a Facebook post that details each waitlist candidate's struggle with ESRD and their need for a live donor. The post is then uploaded to Facebook so it can be shared with the candidate's Facebook social network.
  Interventions: Behavioral: Live Donor Champion + Facebook App
- Facebook App (Active Comparator): The Facebook app provides step-by-step instructions for creating a Facebook post that details each waitlist candidate's struggle with ESRD and their need for a live donor. The post is then uploaded to Facebook so it can be shared with the candidate's Facebook social network. The Facebook App prompts users with specific questions to create a narrative. Links to supplemental resources are auto-populated into the post to provide anyone that views the post with vetted information about the risks, benefits, and process of live donation. Candidates using the Facebook app attend one focus group session held at the transplant center where they are provided with verbal instructions and visual demonstrations of installation and use of the Facebook app.
  Interventions: Behavioral: Facebook App
- Standard of Care (No Intervention): Standard of Care does not include any of the interventions detailed above, but rather normal routine care as this is the control group.

INTERVENTIONS:
Behavioral: Facebook App — This web-based mobile application allows candidates to write a simple and effective story to share with their previously built network on Facebook to help share their story and identify a potential live donor.
  Arms: Facebook App
Behavioral: Live Donor Champion + Facebook App — A "Live Donor Champion" (LDC) is a friend, family member, or community member who serves as an advocate for the candidate in their pursuit of live donation. The investigators have developed a six-month program that provides education and advocacy training to waitlist candidates and their LDCs.
  Arms: Live Donor Champion + Facebook App

SUMMARY:
This pilot study will be a clinical trial to test the feasibility and effectiveness of an educational intervention and a mobile health intervention in adults with end stage renal disease (ESRD) who have not yet identified a potential live donor.

DETAILED DESCRIPTION:
Transplant candidates are hesitant to discuss their illness and the difficulties associated with dialysis, and are therefore reluctant to pursue live donor kidney transplant (LDKT). The investigators will conduct a prospective 3-arm randomized controlled trial with two novel interventions to increase live donation. Arm 1 includes LDC program and the Facebook app, Arm 2 includes just the Facebook app, and Arm 3 includes standard of care. The investigators primary objective is to demonstrate the the effectiveness of these interventions in increasing live donor transplantation rates for candidates with no prior potential live donor.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant candidates aged≥18 added to the waitlist in the last year with no potential live donors are eligible.
* If there is an individual willing to donate, but the candidate is unwilling to consider this option or this particular individual, the candidate is eligible for the trial and may still benefit from identification of new donors or increased comfort accepting donation from others.
* Participants at Johns Hopkins University or University of Alabama must speak English. Participants at Northwestern University must speak English or Spanish.

Exclusion Criteria:

* Candidates with live donors currently under evaluation for donation will be excluded.
* Those with a previous kidney transplant will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 775 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2026-12-07 (Estimated); Study Completion 2026-12-07 (Estimated)

PRIMARY OUTCOMES:
Live donor kidney transplantation | within 1 year of enrollment
  Live donor kidney transplantation within one year of enrollment into the study will be the primary outcome and will be collected/identified through electronic medical record system.

SECONDARY OUTCOMES:
Live Donor Inquiries | within 1 year of enrollment
  Live Donor Inquiries on behalf of candidates will be the secondary outcome and will be collected/identified through electronic medical record system.
knowledge of live donation | within 6 months of enrollment
  knowledge of live donation of transplant candidates will be collected during the survey.
comfort initiating conversations | within 6 months of enrollment
  comfort initiating conversations with others about live donation will be collected during the survey.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Cameron, MD PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Northwestern University, Evanston, Illinois
  - Johns Hopkins University, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No